CLINICAL TRIAL: NCT02056496
Title: Pharmacokinetics and Bioavailability of Pomegranate Phenolics and Gut Microbiota-derived Metabolites (Urolithins) in Overweight Subjects. Comparison Between Two Pomegranate Extracts
Brief Title: Pharmacokinetics and Bioavailability of Pomegranate Phenolics and Urolithins in Healthy Subjects.
Acronym: POMEkinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Full Research Professor, National Research Council, Spain
Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CEBAS-CSIC-3
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Pomegranate; Ellagic acid; Pharmacokinetics; Urolithins; Bioavailability
MeSH Terms: interventions — pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomegranate extract (Experimental): The same group will consume the two types of pomegranate extract (crossover study).
  Interventions: Dietary Supplement: Pomegranate extract

INTERVENTIONS:
Dietary Supplement: Pomegranate extract — Crossover study: The group will consume the pomegranate extract with low punicalagin:EA ratio (PE-1). After 2 weeks of washout, the same group will also consume the other extract with high punicalagin: EA ratio (PE-2).
  Other Names: PE-1
Dietary Supplement: Pomegranate extract — Crossover study: The group will consume the pomegranate extract with high punicalagin:EA ratio (PE-2) after 2 weeks of washout. The same group will also consume the other extract with low punicalagin: EA ratio (PE-1).
  Other Names: PE-2

SUMMARY:
Pomegranate phenolics (such as the ellagitannin punicalagin and ellagic acid) are metabolized by the human gut microbiota to yield a number of metabolites called urolithins (mainly Uro-A). Both ellagic acid (EA) and urolithins can exert a number of biological activities. However, the bioavailability of ellagic acid has been reported to be very low and the existing studies are controversial so far. The investigators want to carry out a robust (cross-over, double-blind) pharmacokinetic assay in 20 healthy volunteers, using two types of pomegranate extracts (PEs). PEs with low (PE-1) and high (PE-2) punicalagin:EA ratio will be administered. The investigators will analyze blood and urine samples using UPLC-ESI-QTOF-MS/MS. The investigators will evaluate:

* The pharmacokinetics of EA.
* The effect of punicalagin:free EA ratio on the pharmacokinetics of EA and urolithins production.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years.
* Healthy status (no illness in the previous 3-months).

Exclusion Criteria:

* Smoking.
* Pregnancy/lactation.
* Severe medical illness/chronic disease/ or gastrointestinal pathology (ulcers, irritable bowel syndrome, ulcerative colitis, Crohn disease etc.).
* Previous gastrointestinal surgery
* Recent use of antibiotics (within 1-month prior to the study)
* Suspected hypersensitivity to pomegranate or any of its components
* Consumption of nutraceuticals, botanical extracts or other vitamin supplements or taking medication.
* Regular consumption of ellagitannin-containing foodstuffs (walnuts, pomegranate, strawberries, raspberries, oak-aged red wine) (after filling a food-frequency questionnaire).
* Intake of ellagitannins-containing foodstuffs the week before the pharmacokinetic intervention.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
24-hour pharmacokinetics of ellagic acid in plasma | Outcome measures at 0.5, 1, 2, 3, 4, 5, 6, and 24 hours post-dose.
  Determination of pharmacokinetic parameters (Cmax, Tmax, AUC, etc.) for ellagic acid and derived metabolites.

SECONDARY OUTCOMES:
72-h accumulation of urolithins in urine | Changes from baseline at 24, 48 and 72 hours
  Production of urolithins depending on the punicalagin:free ellagic acid ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Juan Carlos Espín, PhD, Principal Investigator — National Research Council (CEBAS-CSIC, Murcia, Spain)
Locations (1):
- UCAM (San Antonio Catholic University from Murcia), Murcia, Murcia, Spain